CLINICAL TRIAL: NCT01397110
Title: Influence of Respiratory and Exercise Therapy on Oxygen Uptake, Quality of Life in Patients With Severe Associated Pulmonary Arterial Hypertension (APAH) as Part of a Congenital Heart Defect With / Without Eisenmenger's Syndrome
Brief Title: Respiratory and Physical Therapy in Patients With Associated Pulmonary Arterial Hypertension (APAH) With Congenital Heart Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Ekkehard Gruenig, Prof. Dr. med. Ekkehard Grünig, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011-07-12
Record Dates: First submitted 2011-07-13; First posted 2011-07-19 (Estimated); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Pulmonary Arterial Hypertension; Eisenmenger Syndrome
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Eisenmenger Complex | interventions — Respiratory Rate; Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Respiratory and exercise therapy (Active Comparator): Randomized, prospective, controlled, blinded study of three-week inpatient rehabilitation and subsequent continuing of the training at home for 12 weeks. The control group received conventional rehabilitation without a specific training program. After 15 weeks training is also offered to patients in the control group.
  Interventions: Other: respiratory and exercise therapy
- Control group without exercise training (No Intervention): patients of the control group continue their sedentary lifestyle without given advice for exercise training.
  The time before start of rehabilitation (three months) serves as control group. Afterwards patients take part in the training program as well.

INTERVENTIONS:
Other: respiratory and exercise therapy — Conventional therapy with specific respiratory and physical therapy plus mental walking training
  Arms: Respiratory and exercise therapy

SUMMARY:
The purpose of this study is to investigate the influence of physical training on exercise capacity, quality of life, functional class, oxygen consumption and right ventricular function in patients with severe associated pulmonary arterial hypertension (APAH) as part of a congenital heart defect with / without Eisenmenger's Syndrome

ELIGIBILITY:
Inclusion Criteria:

* signed consent form
* men and women> 18 years <80 years
* APAH with congenital heart defects with / without Eisenmenger syndrome (WHO functional class II-IV), invasively diagnosed by right heart and left heart catheterization: mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg, with targeted PAH medication for at least two months stable before study inclusion (exception: compensated WHO class II without vasodilating drug therapy)

Exclusion Criteria:

* Pregnancy or lactation
* Change in medication during the last 2 months
* severe walking disturbance
* uncertain diagnoses
* No previous invasively confirmation of PH
* acute diseases, infections, fever
* Serious lung disease with FEV1 <50% or TLC <70% of target
* Further exclusion criteria are the following diseases: active myocarditis, unstable angina pectoris, exercise-induced ventricular arrhythmias, recurrent syncope within 4 weeks before study entry

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-01; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the maximum 6-minute walk distance (6MGT) | up to 15 weeks
Changes in quality of life | up to 15 weeks

SECONDARY OUTCOMES:
Changes in hemodynamics | up to 15 weeks
  1. Changes in maximum oxygen uptake
  2. Changes in exercise capacity: 6-minute walk distance, Recumbent Bike (Watts), respiratory economy (EQO2, EQCO2)
  3. Improved condition(NYHA class, Borg scale)
  4. Changes in Magnetic resonance tomography and echocardiographic parameters of right and left ventricle: size and pump function.
  5. Change of laboratory parameters, which are markers of right heart failure as NTproBNP, interleukins

CONTACTS AND LOCATIONS:
Overall Officials: Ekkehard Gruenig, MD, Study Chair — Center for pulmonary hypertension, Thoraxclinic Heidelberg
Locations (1):
- : Center for pulmonary Hypertension, Thoraxclinic Heidelberg, Heidelberg, Germany